CLINICAL TRIAL: NCT01724255
Title: The Influence of the Timing of Staple and Dressing Removal After Cesarean Section on the Surgical Incision Healing
Brief Title: Optimal Time for Staple/Dressing Removal
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: StapleDressingRemoval-HMO-CTIL
Record Dates: First submitted 2012-11-07; First posted 2012-11-09 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Surgical Wound Healing; Surgical Wound Infection; Patient Satisfaction
Keywords: Caesarian section; Surgical Wound
MeSH Terms: conditions — Surgical Wound Infection; Patient Satisfaction; Surgical Wound | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- staple removal day 4 dressing removal day 1: early staple removal and early dressing removal
  Interventions: Other: questionnaire
- staple removal day 4 dressing removal day 4: early staple removal and day 4 dressing removal
  Interventions: Other: questionnaire
- staple removal day 7, dressing removal day 1: late staple removal and early dressing removal
  Interventions: Other: questionnaire
- staple removal day 7, dressing removal day 7: late staple removal and late dressing removal
  Interventions: Other: questionnaire
- staple removal day 7, dressing removal day 4: late staple removal and day 4 dressing removal
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire

SUMMARY:
The medical literature does not provide sufficient information or recommendation regarding the optimal time to remove the staples and the bandage after a cesarean section. The goal of this study is to compare 5 groups of patients:

1. staple removal on POD 4 and dressing removal on Post Operative Day (POD)1
2. staple removal on POD 4 and dressing removal on Post Operative Day (POD)4
3. staple removal on POD 7 and dressing removal on Post Operative Day (POD)1
4. staple removal on POD 7 and dressing removal on Post Operative Day (POD)7
5. staple removal on POD 4 and dressing removal on Post Operative Day (POD)7

Since there is no definite protocol for staple and dressing removal, we will adapt the above protocol each for a 3-4 month period of time. Patients will be contacted to either return for a follow up visit or to answer a telephone survey.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing a cesarean section at our facility

Exclusion Criteria:

* patients lost to follow up

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients undergoing a cesarean section at our facility
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Wound infection and complications | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Drorith Hochner-Celnikier, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Heinemann N, Solnica A, Abdelkader R, Gutman J, Nalbandian N, Raizman E, Hochner-Celnikier D. Timing of staples and dressing removal after cesarean delivery (the SCARR study). Int J Gynaecol Obstet. 2019 Mar;144(3):283-289. doi: 10.1002/ijgo.12757. Epub 2019 Jan 11. PMID 30582610